CLINICAL TRIAL: NCT03471390
Title: Identification and Development of Interfaces and Processes to Improve Quality of Life of Residents at Senevita ProQuaS 2- Improving Pain Management in Nursing Homes: a Pilot Study
Brief Title: Improving Pain Management in Nursing Homes: a Pilot Study
Acronym: ProQuaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: Senevita AG (Unknown)
Responsible Party: Principal Investigator, Franziska Zúñiga, University lecturer, University of Basel
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: ProQuaS
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Pain Management
Keywords: Nursing Home
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: non- randomized incomplete stepped-wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ProQuaS 2- Intervention (Experimental)
  Interventions: Other: ProQuaS 2 Intervention

INTERVENTIONS:
Other: ProQuaS 2 Intervention — Training and implementation of facility pain champions, comprehensive training of all care workers in pain assessment and management, implementation of pain management policies

SUMMARY:
This study aims to improve pain management in Swiss nursing homes by addressing behavior change of the care workers with a multilevel intervention

DETAILED DESCRIPTION:
Pain management in nursing homes often is inadequate despite the availability of evidence- based pain management guidelines. Barriers to pain management in nursing homes occur on several levels including lack of knowledge and negative beliefs towards pain of care workers.

For this embedded mixed-methods pilot study a convenience sample of maximum six nursing homes will be recruited. The planned intervention comprises the implementation of pain management policies, training of all care workers in pain assessment and management as well as training and introduction of a facility pain champion. Quantitative outcomes assessed at baseline, after three and six months include self-efficacy and attitudes to pain of care workers, functional interference from pain and pain intensity in residents. Feasibility and acceptability of the intervention and potential barriers to its implementation will be explored in focus groups and interviews.

ELIGIBILITY:
Inclusion Criteria:

Care workers:

* Registered nurses, licensed practical nurses/certified caregivers, nursing assistants, nurse aides and other care workers from the participating nursing home
* Working in direct resident care
* Participating care workers have to be employed for at least one month at the data collection
* Students, apprentices and interns have to be employed at least six months in total
* Speak and understand German
* Older than 16 years

Residents:

* All residents living in a participating nursing home, older than 64 years
* Written informed consent to participate in data collection signed by the resident or in case of severe cognitive impairment by his/her legally acceptable representative

Exclusion Criteria:

Care workers:

* Temporary employment for less than six months

Residents:

* Critical current health status or terminal life situation
* Known life expectancy less than 3 months
* Short term residents (length of stay <6 months)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Self- efficacy in pain management | Change from baseline to 6 months
  Care workers' self-efficacy in pain management scale
  * investigator-developed scale based on guide for constructing self-efficacy scales (Bandura 2006)
  * numeric rating scale ranging from 0 ="not confident at all" to 100="highly confident"
  * total score will be computed by calculating a mean over single item scores (range: 0-100, higher scores indicating better self-efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Zúñiga, PhD, Principal Investigator — University of Basel
Locations (4):
- Switzerland (4):
  - Senevita Obstgarten, Affoltern am Albis
  - Senevita Gellertblick, Basel
  - Senevita Wangenmatt, Bern
  - Senevita Aespliz, Ittigen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunkert T, Ruppen W, Simon M, Zuniga F. A theory-based hybrid II implementation intervention to improve pain management in Swiss nursing homes: A mixed-methods study protocol. J Adv Nurs. 2019 Feb;75(2):432-442. doi: 10.1111/jan.13817. Epub 2018 Sep 6. PMID 30109728